CLINICAL TRIAL: NCT00202241
Title: The Effects of Anabolic Steroids and Protease Inhibitors on Serum Blood Lipids,Muscle Mass, and Total Body Fat in People Living With HIV/AIDS
Brief Title: The Effects of Anabolic Steroids and Protease Inhibitors on People Living With HIV/AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Dr. Wendy Wobeser, Principal Investigator, Queen's University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DMED-99
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: HIV; AIDS; Lipodystrophy; Hyperlipidemia
Keywords: HIV; AIDS; testosterone; anabolic steroid; body composition; lipodystrophy; MRI; BIA; skinfold measurements; protease inhibitors
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Lipodystrophy; Hyperlipidemias | interventions — Testosterone

INTERVENTIONS:
Procedure: testosterone injection

SUMMARY:
The main aim of the study is to investigate the combined effects of using anabolic steroids and protease inhibitors on fat metabolism and body composition of People Living with HIV/AIDS.

We are seeking to answer the following questions:

1) Are there any significant differences in serum blood lipids, lipodystrophy, in persons with HIV taking antiretroviral therapies and anabolic steroids versus antiretroviral therapies alone?

DETAILED DESCRIPTION:
Changes in body composition and wasting have been a constant concern for people living with HIV/AIDS. Testosterone and its derivatives, anabolic steroids (AS) are being used by persons with HIV/AIDS (PHA's) to treat AIDs related wasting syndrome and also for bodybuilding purposes. some studies have shown that AS had a positive impact on the weight and well-being of HIV seropositive individuals.

It has been shown that protease inhibitors (PI's) in combination with other antiretroviral HIV therapies are associated with a symmetrical loss of subcutaneous fat from the body surface (lipodystrophy)in some PHAs.

The mechanism for lipodystrophy is not well understood. However, it is associated with hyperlipidemia that contributes to central fat deposition, insulin resistance, and in some, type 2 diabetes. As well, increased visceral abdominal fat and loss of fat inthe arms, legs and face, and increased levels of serum lipids have been reported.The health effects of anabolic steroid therapy coupled with PIs has not been examined before.

This study is an observational study investigating the phenomenon of lipodystrophy in an HIV population already exposed to AS and PIs. A prospective observational design will be employed, with two groups recruited. One group will be taking AS and PI's, the other will be taking PIs only.

The groups will be asked to completed Quality of Life nutrition and physical activity questionnaires. Serum blood lipid characteristics will be compared, and body composition will be determined using MRIs, BIA's and skinfold measurements.

ELIGIBILITY:
Inclusion Criteria:

* documented HIV seropositive status
* 18 years of age or older
* combination antiretroviral therapies for at least three months or more
* able to comply with study procedures and protocol
* signed informed consent

Exclusion Criteria:

* acute opportunistic infections at baseline
* use of serum lipid lowering drugs
* use of serum sugar controlling drugs
* evidence of drug or alcohol use which may interfere with study participation
* a recent illness with associate weight loss of greater than or equal to 10lbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 1999-09; Study Completion 2001-06

PRIMARY OUTCOMES:
differences in serum lipid levels
differences in regional and overall body fat level
impacts on metabolic and cardiovascular health

SECONDARY OUTCOMES:
quantity of muscle tissue between group comparison
comparison of 3 determinants of body composition(MRI,skinfold,BIA)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Wobeser, MD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada